CLINICAL TRIAL: NCT07110623
Title: Real-time Molecular Diagnosis of Oral Precancer
Acronym: LIP
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 307234; 307234 (Other: Health Research Authority (HRA) UK)
Record Dates: First submitted 2025-07-08; First posted 2025-08-07 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Oral Cancer; Dysplasia; Oral Lesions; Oral Pre-cancer; Mouth Cancer
Keywords: oral cancer; mouth lesions; dysplastic oral lesions; mouth cancer; pre-cancer; mouth pre-cancer; oral pre-cancer; oral lesions; oral biopsy; polarized Raman spectroscopy
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient group: 1. Has a medical condition for which biopsy of oral tissue has been indicated.
  2. Is undergoing inspection for early oral cancer
  Interventions: Device: LIP device
- Healthy controls: Participants who have healthy oral tissue
  Interventions: Device: LIP device

INTERVENTIONS:
Device: LIP device — The LIP device uses polarized Raman spectroscopy to enhance the early detection and diagnosis of oral cancer by facilitating more accurate guiding of biopsies. This non-invasive technology utilizes polarized laser light to generate Raman scattering that can be used to analyze molecular vibrations, which in the future will provide clinicians with insights into tissue composition and structure for identifying cancerous abnormalities.

SUMMARY:
The "Real-time molecular diagnosis of oral precancer" or the LIP study is testing a new device for the detection of cancer in the mouth.

Oral cancers are serious and devastating illnesses, especially if detected at a late stage. Currently, the detection of oral cancer relies on testing a biopsy, which involves cutting a small section of tissue from the mouth and sending it to the pathology laboratory for further testing. A doctor or dentist taking the biopsy must rely on their own eyesight and experience to spot areas of concern. It can therefore be difficult to detect the earliest stages of cancer. At times, cancer tissue is only detected because it has already developed, and this affects the success of the treatment.

The device tested in this study uses a laser beam to scan areas inside the mouth and a computer collects information about the scan. The goal of this project is to train the computer software in the device to recognize pre-cancer and cancer from normal scans. Patients who need to have a biopsy due to suspected pre-cancer or cancer in the mouth will be scanned with the device. Biopsy reports will be used to tell the software which scans were from pre-cancer or cancer or non-cancer tissues. Volunteers with healthy oral tissue will be included to further test the computer software. Secondary aims include collecting pilot safety data and feedback regarding the use of this device. If successful, the results from this pilot study will lead to a bigger trial to further study how the device can be used for cancer diagnosis.

DETAILED DESCRIPTION:
Oral cancers are severe life-limiting diseases, particularly when diagnosed in late stages. Earliest possible detection in precancer (dysplasia) or early cancer stages is the single most important measure for reducing oral cancer patients' morbidity and mortality rates. Conventional diagnosis relies on visual inspection guiding the biopsy of suspicious oral lesions, which has resulted in 5-year survivals of up to 90% for early tumors or dysplasia. This survival rate however declines to at best 50% for advanced cancers, highlighting the necessity of early diagnosis as a primary factor in determining patient outcomes. Visually guided tissue sampling suffers from inter-observer dependence, sampling errors and difficulty in identifying and targeting flat dysplastic lesions in particular. The differentiation between inflamed/scarred tissue and dysplasia, establishing cancer depth, local/distant spread assessment (staging) and grading (aggression), and margin assessment of malignant lesions, all represent monumental clinical challenges. Further, biopsy also remains a significant deterrent to patient attendance. There is a significant unmet clinical need for a rapid, non-invasive, outpatient-deployable diagnostic method to improve surveillance, early diagnosis, and follow up / management of oral cancer patients.

Optical imaging and spectroscopy have recently offered great promise to address unmet clinical needs since they are non-invasive and can capture molecular/structural information without prior tissue preparation. These technologies offer new, clinically relevant biomarkers such that essential point-of-care decisions can be made with the use of safe (non-ionizing) levels of optical radiation at a much lower cost than with MRI, CT and PET. Raman spectroscopy is a label-free, rapid and minimally invasive optical technique using laser light that provides a point-wise optical fingerprint of the myriad of inter- and intra-cellular building blocks of tissue (i.e., proteins, lipids and DNA) at the biomolecular level. Raman spectroscopy offers label-free diagnosis of cancers in vivo. In the last two decades, there has been accumulating evidence on the accurate diagnostic capability of Raman spectroscopy through comprehensive in vitro, ex vivo and in vivo studies.

The research team have developed a 2nd generation polarized Raman platform that provides polarized Raman signals and is compatible with the oral cavity. It can provide a point-wise vibrational molecular fingerprint "optical biopsy" of both tissue structure/molecular symmetries and composition. The key advantage of polarized Raman spectroscopy compared to conventional Raman spectroscopy is that it offers additional specific information about tissue structure and organization. The developed prototype is fully functional and will allow us to take the first step towards translation of the developed clinical platform technology.

In this study, patients with suspected pre-cancer or being seen by a clinician for early oral cancer will be recruited. The participants will be scanned with the LIP device and will have a biopsy if this was planned as part of their routine care. Health volunteers will be recruited to increase the number scans of healthy tissue and to help validate the device. The primary aim of this study is to collect the output of the scans and train the device to discriminate premalignant/malignant conditions from benign oral tissue. No clinical output will be provided at this stage, thus diagnosis of suspicious lesions will be confirmed through a biopsy according to standard NHS procedures. Secondary aims include collecting pilot safety data, and feedback from users of the device and study participants.

ELIGIBILITY:
Inclusion criteria for patients

1. Adult aged 18 and older
2. One of the following criteria must be met:

   1. Has a medical condition for which biopsy of oral tissue has been indicated.
   2. Is undergoing inspection for early oral cancer
3. Willing and able to comply with all study procedures.

Exclusion criteria for patients

1. Has a bleeding disorder, such as haemophilia, or has contraindication for having a biopsy.
2. Severe co-morbid illness, such as end-stage renal failure (ESRF), congestive cardiac failure (CCF), severe osteoarthritis (OA) and rheumatoid arthritis (RA) requiring long term non-steroidal anti-inflammatory drug (NSAID) therapy and any other immunosuppression / immuno-modulation therapy.
3. Has other severe acute or chronic medical or psychiatric condition where use of the device may cause unnecessary stress
4. Any condition that under judgment of the investigator would make the subject unsuitable as it may interfere with interpretation of study results
5. Currently using any compound recognised as acting as a light sensitizer / has a recognised condition associated with light sensitisation / tissue sensitivity to light such as photodynamic therapy or lupus.
6. Is pregnant or breastfeeding
7. Has a laboratory abnormality in medical record that may interfere with the interpretation of study results

Inclusion criteria for healthy volunteers

1. Adult aged 18 and older.
2. Willing and able to comply with all study procedures.

Exclusion criteria for healthy volunteers

1. Has a medical condition for which biopsy has been indicated or is undergoing inspection for early cancer.
2. Severe co-morbid illness, such as end-stage renal failure (ESRF), congestive cardiac failure (CCF), severe osteoarthritis (OA) and rheumatoid arthritis (RA) requiring long term non-steroidal anti-inflammatory drug (NSAID) therapy and any other immunosuppression / immuno-modulation therapy.
3. Has other severe acute or chronic medical or psychiatric condition where use of the device may cause unnecessary stress
4. Any condition that under judgment of the investigator would make the subject unsuitable as it may interfere with interpretation of study results
5. Currently using any compound recognised as acting as a light sensitizer / has a recognised condition associated with light sensitisation / tissue sensitivity to light such as photodynamic therapy or lupus.
6. Is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from a single site at Guy's Hospital (London, UK).
  Patients with suspected pre-malignant or malignant condition (ie. having a "suspicious lesion") will be recruited from oral medicine and dental clinics at Guy's Hospital (London, UK) during their hospital appointment.
  Healthy volunteers will be recruited from staff and students at KCL and GSTT.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the collection of spectra from the oral cavity of each participant, including premalignant, malignant lesions and benign tissues within the same individuals. | Day 1
  Spectra outputs from the device will be collected from the device computer and matched to biopsy results for patients enrolling in the study. For healthy controls, spectra will be collected and assigned as being scanned from healthy tissue.

SECONDARY OUTCOMES:
Pilot safety data collected through adverse events monitoring | From the point of scan up to 24 hours after the device scan
  Pilot safety data will be collected for study participants and users of the device by recording adverse events from participants after the scan and from device users when using the scan.
Participant feedback about having a scan with the LIP device using bespoke questionnaire | Day 1
  Feedback from study participants will be collected regarding their experience of having an oral scan with the LIP device. The "LIP Feedback Questionnaire for participants" was designed specifically for this study to capture feedback through Likert-type questions and free text boxes. Answers are not reported using a scale.
User acceptability and feedback about the LIP device using bespoke questionnaire | Day 1
  To better understand the experience of users of the device, feedback will be collected on the "LIP Feedback Questionnaire for users of the device" which was created to capture the device user experience with Likert-type questions and free text boxes. Answers are not reported using a scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mads Bergholt, PhD, Study Chair — King's College London; Richard J Cook, PhD, MRCSEd, MBChB, FDS RCS, Principal Investigator — King's College London
Locations (1):
- Oral Clinical Research Unit, Guy's Hospital, London, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No